# Research Protocol SUMMARY.version 8.7.2024

Study Title: Baclofen as a Perioperative Analgesic Adjuvant for Kidney Stone Surgery

Principal Investigator: Mark Mandabach MD

First subject studied: 10/27/2020 Final subject studied: 10/27/2022

Original IRB Approval Date: April 12, 2019

Modifications of Consent forms to final REDCap version utilized in enrollment: August 2, 2019

Published: Mandabach M, Deichmann P, Massoll A, Graves S, Assimos D, Wood K and Ness TJ. Use of baclofen premedication as an analgesic adjuvant in patients undergoing percutaneous nephrolithotripsy: a placebo-controlled, double-blind randomized trial. *Cureus* DOI: 10.7759/cureus

| INDEX | <u>Section</u> |
|--------------------------------|----------------|
| Summary of Study | 1.0 |
| Background & Rationale | 2.0 |
| Objective(s) & Hypothesis | 3.0 |
| Inclusion & Exclusion Criteria | 4.0 |
| Randomization Procedures | 5.0 |
| Study Interventions/Procedures | 6.0 |
| Plan for Study | 7.0 |
| Drug and Device Information | 8.0 |
| Statistical Considerations | 9.0 |
| References | 10.0 |

#### 1.0 **SUMMARY OF STUDY**

The present study proposes to study the effect of a single preoperative dose of baclofen on pain treated in the first 24 hours after kidney stone-related surgeries using a placebo-controlled, double-blind methodology. Because this patient population often has a history of significant opioid use, which would be expected to alter postoperative pain medication requirements, patients will be stratified into those which would be expected to be opioid tolerant (use >30 OME daily) and those who are generally opioid naïve.

## 2.0 BACKGROUND & RATIONALE

Postoperative pain continues to be a significant clinical problem. Use of perioperative adjuvants has improved postoperative pain control. The GABA-B receptor agonist, baclofen, is an appropriate drug to trial as such an analgesic adjuvant. Support for this assertion is given below

**Baclofen pharmacology.** The drug baclofen (chemical name) is a GABA derivative. Its mechanisms of action is through the metabotropic GABA-B receptor and is G-protein linked to potassium channels leading to neuronal hyperpolarization. Baclofen is a white powder, practically odorless powder which is manufactured in 10 and 20 mg tablets with typical doses for spasticity of 10-20 TID. It is rapidly absorbed and has half-life of 2-4 hours. 85% of the compound is excreted unchanged in urine.

Sites of action are peripheral, spinal and supraspinal. Selective spinal infusion is utilized to control spasticity. Notable for this discussion, CASL imaging of the brain before and after 21 days of baclofen treatment (20 QID) demonstrated reduced rCBF in the ventral striatum and medial prefrontal cortex and increased rCBF in the lateral OFC, (a region involved in suppressing previously rewarded behavior) and cerebellum. rCBF was also blunted in the insula bilaterally [Franklin et al, 2011].

Baclofen produces analgesia. Baclofen produces analgesia by itself as measured in rats and mice in the hot plate, tail flick and acetic acid-induced writhing [Aley and Kulkarni, 1989, 1991; Balerio and Rubio; mult other] In rats with chronically inflamed paws baclofen increased Substance P release raising issues related to acute vs. chronic analgesic benefits of the GABA-B agonists [Malcangio and Bowery, 1994; Galeotti et al 1996]. Baclofen produced analgesia in primates in the formalin test [Sharma et al, 1993]. In chemotherapy-induced neuropathic pain models baclofen produced significant but erratic analgesia [Xiao et al, 2008]. Intrathecal nociceptin antagonized baclofen-induced analgesia in a mouse tail flick assay [Citterio et al, 2000] and baclofen-induced analgesia was absent in GIRK2 knockout mice [Blednov et al] Baclofen administered spinally (intrathecally) produces analgesia in rat thermal pain models that can be antagonized by GABA-B antagonists [Aran and Hammond]. Whitehead et al [2012] demonstrated peripheral analgesic effects of baclofen in a mouse arthritis model.

Baclofen's analgesic effects may be acting via the same mechanism by which heterosegmenal noxious stimuli produce inhibition (nocigenic inhibition) since such inhibition has been demonstrated to act via GABA-B and mu opioid mechanisms [Tambell et al, 2009]. Consistent with this, analgesia produced by 100 Hz electroacupuncture as involves GABA-B mechanisms [Silva et al]. GABA-B receptor blockade also blocks foot-shock induced "stress-induced" analgesia, but not forced swim stress or psychological stress [Tokuyama et al] although others have observed potentiation of forced swim stress-induced analgesia by baclofen [Houston et al, 1997]. In the spinal substantia gelatinosa activation of GABA-B receptors presynaptically block neurotransmitter release [Yang and Ma] and NK1 receptor expression [Enna et al]. Other sites of action related to pain include the rostral agranular insular cortex [Jasmin et al] and lateral preoptic area [Lim et al]. The supraspinal analgesic effects of baclofen appear to act via adrenergic and opioidergic spinal mechanisms [Jasmin et al; Ignatov and Andreev;] with potentially a cholinergic and GABA-A portion to contribution [Tamayo et al 1988; Zarridast MR and Djavdan M].

In humans, baclofen has had a particular role as an anesthetic for cranial nerve-related neuropathic pains such as trigeminal neuralgia [Knotkova and Pappagallo]. Early anecdotal reports (e.g. Harmer and Larson) suggested it worked for postherpetic neuralgia in facial distributions but not spinal distributions [Terrence et al, 1985]. In humans, the spinal administration of baclofen has also demonstrated short-term analgesic effects on spinal cored injury-related pain and post-stroke pain [Taira et al, 1995]. One presumed mechanism for the action of baclofen on facial pain is the presence of GABA-B receptors on

trigeminal primary afferent neurons whose activation leads to a potentiation of voltage-dependent potassium currents. Baclofen has demonstrated analgesic effects on surgical pain in females [Corli et al]

**Baclofen interacts with opioids synergistically.** Gordon et al (1995) observed potentiation of morphine analgesia on post-operative pain but not of pentazocine-induced (kappa) analgesia. Panerai et al [1985] had previously demonstrated baclofen prolonged the analgesic effect of fentanyl on post-operative pain. Notably, baclofen also potentiates the analgesia produced by clonidine in rat models [Przesmycki et al]

**Baclofen reduces addictive behaviors.** In a randomized, double-blind placebo-controlled clinical trial Assadi et al [2003] used baclofen for the maintenance treatment of opioid dependence. In a 12 week trial of 20 TID. Baclofen was superior over placebo in terms of opiate withdrawal syndrome and depressive symptoms. Trends towards reductions in opioid craving and self-reported opioid and alcohol use were noted but not proven.

Baclofen has also been noted to reduce cigarette consumption [Franklin et al, 2009]

Corwin et al [2012] in a double-blind, placebo-controlled, crossover study in 12 subjects demonstrated that baclofen (20 TID) reduced binge-eating. Slight but significant increases in depression symptomatology occurred. Tiredness, fatigue and upset stomach were the most commonly reported side effects.

Ling and Shoptaw [1998] in a clinical series of ten patients reported reduced cocaine-craving due to baclofen with good safety and tolerability. General reviewes posit its beneficial effects in multiple forms of addiction [Kumar et al, 2013]

The place in the treatment of addictive behaviors where baclofen treatment has found its greatest audience is in the realm of alcohol addiction [reviewe – Gorsane et al] but with mixed results for efficacy by placebo-controlled, double-blind randomized trials [e.g. Garbutt et al 2010]. Effects on alcohol craving, use and abuse have also been demonstrated with general acceptance of beneficial effects but varying levels of effect [Dore et al, 2011; Vuittonet et al 2014; Tyacke et al, 2010; Leggio et al, 2010; Johnson et al, 2005] – similar benefits have been noted for GABA-B positive allosteric modulators [Filip et al, 2014]

Baclofen reversed cognitive deficits induced by acute cocaine in rhesus monkeys and normalized activation of prefrontal cortex sites[Porrino et al, 2014]

In rat models, baclofen dose-dependently reduced heroin-seeking behavior [Spano et al, 2007], reversed behavioral sensitization to morphine [Bartoletti et al, 2007] and prevents heroin-induced reinstatement of heroin-seeking behaviors [Spano et al, 2007] and enhances extinction of opiate and methamphetamine-induced conditioned place preference [Heinrichs et al, 2010; Voigt et al, 2011] particularly stress-accenuated morphine-induced conditioned place preference [Meng et al, 2014]. In rodent models of cocaine- or heroin-seeking behaviors, baclofen was found to attenuate these behaviors [DiCiano and Everitt, 2003]. Similar results are noted for alcohol-seeking and drinking behavior [Maccioni and Colombo, 2009].

Baclofen reduced ethanol consumption in mice, but only in those which were phenotypically less prone to heavy drinking behaviors [Villas Boas et al, 2012]. Baclofen reduced nicotine- [Paterson et al, 2004] and morphine self-administration in rats and a GABA(B)-antagonist increased morphine administration [Ramishini et al, 2013]

Baclofen administered into the locus coeruleus attenuated morphine withdrawal signs [Riahi et al, 2009]

Presumed mechanisms for baclofen's actions on addictive behaviors is an interaction wth dopaminergic neurons of the ventral tegmental area where baclofen leads to Girk signaling [Arora et al, 2011] with a subsequent reduction in dopamine release in the nucleus accumbens.

Baclofen toxicology and drug/drug interactions. There have been limited toxicities or side effects of baclofen. Odd reactions include things such as the induction of hiccup-like respirations [Srivasta et al, 2014] or diabetes insipidus [Silversides and Scott] In rats, intraventricular baclofen impaired memory [Zarrindast et al, 2001] CB1 receptor antagonism decreases analgesia due to baclofen and GABA(B) antagonists reduce analgesia due to cannabinoids [Naderi et al, 2005].

Most toxicity reports relate to withdrawal [Ross et al, 2011] or excessive dosing [Roy and Wakefield, 1986; Leung et al2006] with CNS effects predominant (loss of consciousness, delirium, hypertension). Because it is kidney-cleared, toxicity is more common in patients with advanced nephropathy [El-Husseini et al, 2011]

Some increases in depression have been noted, but in the spinal cord injury patients, use of baclofen improved psychiatric symptoms [Margetis et al, 2014]

DeFeudis [1984] suggested that GABAergic drugs might have a role in both analgesia and drug addictions, particularly related to opioids but did not go so far as to suggest co-administration.

#### 3.0 **OBJECTIVE(S) & HYPOTHESIS**

Purpose of study:

To determine whether a single, oral dose of baclofen alters postoperative opioid requirements

Study Hypothesis:

We hypothesized that a single, oral dose of baclofen given to patients undergoing kidney stone surgery will reduce postoperative opioid requirements measured in the PACU and in the first 24 hours following surgery.

#### 4.0 **INCLUSION & EXCLUSION CRITERIA**

Inclusion criteria:

Adult patients (age >= 19 y.o.) scheduled for kidney stone-related surgery

Exclusion criteria:

[1] History of allergy to baclofen [2] Any condition which might limit appropriate report and treatment of postoperative pain (e.g., non-English speaking; severe psychiatric disease)

# 5.0 RANDOMIZATION/RECRUITMENT DETAILS (If applicable)

Randomization groups, how will subjects be randomized:

All subjects who are patients of Drs. Assimos and/or Wood and scheduled for kidney stone-related surgery will be potentially recruited.

Part 1: In an initial open run-in period, six patients will be recruited and given a dose of 10 mg baclofen preoperatively so that potential side effects can be assessed in an unblinded fashion.

Part 2: After that, patients will be identified and initially stratified into two groups based on preoperative opioid use. If daily using >30 Oral Morphine Equivalents (OMEs) for more than one month they will be designated as Opioid Tolerant. Otherwise, they will be included in the Opioid Naïve group. These two groups will then be each randomized (envelope assignment) into receiving either baclofen (10 mg, p.o. x 1) or placebo as a preoperative medication such that there will be 4 groups of 20 patients identified:

Group 1: Opioid Tolerant - baclofen

Group 2: Opioid Tolerant – placebo

Group 3: Opioid Naïve - baclofen

Group 4: Opioid Naïve - placebo

Blinded 

☐ Yes ☐ No (Single ☐ Double ☐ please check box).

#### 6.0 **STUDY INTERVENTIONS/PROCEDURES**

Study design: Placebo-controlled double-blind

Comparison groups (for prospective and clinical trials only).

Placebo treated individuals

Timeline of interventions (for prospective and clinical trials only).

Patients will be recruited preoperatively by Drs. Assimos and Wood, in addition to anesthesiology-related personnel in the KPAC. Informed consent will be obtained at that time. On the Day of Surgery, subjects will be contacted by study personnel in the Preoperative Holding area to confirm patient participation and then a randomization envelope containing a single dose of either baclofen or placebo will be opened (Groups 1&2 intermixed; Groups 3&4 intermixed; envelopes will be prepared ahead of time by a different investigator according to a randomization table). Subjects will then consume the pill in the envelope and this will be recorded. Patients will then be treated intraoperatively and postoperatively according to the standard of care associated with these surgeries but with an attempt to utilize consistent doses of intraoperative opioids other agents across groups and standardized PACU orders. After discharge from the

PACU patients' pain will be treated with PCA morphine. Notably, the treating anesthesiologist and all PACU personnel will be blinded to the drug that was administered preoperatively. The total use of analgesics, measures of any other side effects (nausea, excessive sedation) will be recorded for 24 hours.

#### Measured Outcomes:

- a. Primary outcomes: Postoperative opioid consumption (measured as OMEs)
- b. Secondary outcomes: Incidence of nausea/vomiting; excessive sedation per patient self assessment; any other untoward events

### 7.0 PLAN FOR STUDY: Click here to enter text.

- a. What is the potential impact of your study findings (e.g., how will findings impact clinical outcomes)? Baclofen may prove beneficial as a perioperative analgesic adjuvant the long term goal would be to determine potential efficacy, safety and tolerability of baclofen use and to perform a follow-up study in which baclofen would be co-administered postoperatively for up to 2 weeks. The conversion from acute to chronic pain and the potential anti-reward effects produced by baclofen could impact subsequent opioid use and abuse.
- b. Do you plan to submit an abstract based on this project? ⊠ Yes ☐ No (If yes, to which meeting venue? Click here to enter text.
- c. Do you intend to publish the finding from this research project:  $\boxtimes$  Yes  $\square$  No

# 8.0 **DRUG INFORMATION**

<u>Drug Name</u>: baclofen hydrochloride

Classification: Antispastic; GABA-B receptor agonist

Mode of Action: GABA-B receptor agonist

Storage and Stability: Pharmacologically stable

Metabolism: Cleared unchanged through kidneys; half-life 2-4 hours

Preparation: Pill

Administration: Oral

Incompatibilities: None

- Contraindications: allergy to baclofen
- Precautions: very safe medication with long track record of clinical use

Click here to enter text.

**Side Effects:** Adverse effects indicated in *italics* are the most frequent adverse effects. Adverse events in bold are severe/life-threatening, otherwise they are mild to moderate in reaction.

CNS: sedation, mild

CV: no major

**EENT**: no major

ENDO: no major

GI: no major

GU: no major

INTEG: no major

MS: weakness at excessive doses

Investigational New Drug (IND) Application required (check yes or no): ☐Yes ☐No

## 9.0 STATISTICAL CONSIDERATIONS

 Original Plan for Statistical Analysis: Data analysis will be by ANOVA analysis using Tukey's HSD for post-hoc analysis for primary outcome data and Fishers Exact test for categorical incidence data. A mid-point analysis was proposed after the study of 40 subjects.

#### 10.0 REFERENCES

- Aley KO and Kulkarni SK. GABAergic agents-induced antinociceptive effect in mice.. Methods Find Exp Clin Pharmcol. 1989 11: 597-601
- 2. Aley KO and Kulkarni SK. Baclofen analgesia in mice: a GABA B mediated mechanism. Methods Find Exp Clin Pharmcol. 1991 13: 681-686
- 3. Aran S and Hammond DL. Antagonisms of baclofen-induced antinociception by intrathecal administration of phaclofen or 2-hydroxy-saclofen, but not  $\delta$ -aminovaleric acid in the rat. J. Pharm Exp Ther 257: 360-368, 1991
- Arora D, hearing M, Haluk DM, Mirkovic K, Fajardo-Serrano A, Wessendorf MW, Watanabe M, Lujan R and Wickman K. Acute cocaine exposure weakens GABA-B receptor-dependent Girk signaling in dopamine neurons of the ventral tegmental area. J. Neurosci 31: 12251-12257, 2011
- 5. Assadi SM, Radgoodarzi R and Ahmadi-Abhari S. Baclofen for maintenance treatment of opioid dependence: a randomized double-blind placebo-controlled clinical t rial. BMC Psychiatry 3:16, 2003.
- 6. Balerio GN and Rubio MC Baclofen analgesia: involvement of the GABAergic system. Pharmacol Res. 46: 281-286, 2002.

- 7. Bartoletti M, Ricci F and Gaiardi M. A GABA(B) agonist reverses the behavioral sensitization to morphine in rats. Psychopharmacol.(Berl) 192: 79-85, 2007.
- 8. Blednov YA, Stoffel M, Alva H, Harris RA. A pervasive mechanism for analgesia: activation of GIRK2 channels. PNAS 100: 277-282, 2003
- 9. Butler SF, Budman SH, Fernandez KC Houle B, Benoit C, Katz N and Jamison RN. Development and validation of the Current Opioid Misuse Measure. Pain 130:144-156, 2007
- 10. Citterio F, Corrandini L, Smith RD and Bertorelli R. Nociceptin attenuates opioid and GABA-B receptor-mediated analgesia in the mouse tail-flick assay. Neurosci Letts 292: 83-86, 2000.
- 11. Corli O, Roma G, Bacchini M, Battagliarin G, DiPiazza D, Brambilla C, Grossi E. Double-blind placebo-controlled trial of baclofen, alone and in combination, in patients undergoing voluntary abortion. Clin Ther 6: 800-807, 1984.
- 12. Corwin RL, Boan J, Peters KF and Ulbrecht JS. Baclofen reduces binge eating in a double-blind, placebo-controlled, crossover study. Behav Pharmacol 23: 616-625, 2012
- 13. Crana SE and Fudin J. Drug interactions among HIV patients receiving concurrent antiretroviral and pain therapy. Practical Pain Management 11:1 (www.practicalpainmanagement.com)
- 14. DeFeudis FV. GABAergic analgesia: implications for GABAerigic therapy for drug addictions Drug Alcohol Depend 14: 101-111, 1984.
- 15. DiCiano P and Everitt BJ. The GABA-B receptor agonist baclofen attenuates cocaine- and heroin-seeking behavior by rats. Neuropsychopharmcol 28: 510-518, 2003.
- Dore GM, Lo K, Juckes L, Bezyan S., Latt N. Clinical experience with baclofen in the management of alcohol dependent patients with psychiatric comorbidity: a selected case series. Alcohol Alcohol 46: 714-720, 2011.
- 17. El-Husseini A, Sabucedo A, Lamarche J, Courville C and Peguero A. Baclofen toxicity in patients with advanced nephropathy: proposal for new labeling. Am J Nephrol 34: 491-495, 2011
- 18. Enna SJ, Harstad EB, McCarson KE. Regulation of neurkinin-1 receptor expression by GABA(B) receptor agonists. Life Sci. 62: 1525-1530, 1998.
- 19. Fadda P., Scherma M, Fresu A, Collu M and Fratta W. Baclofen antagonizes nicotine-, cocaine- and morphine-induced dopamine release in the nucleus accumbens of rat. Synapse 50: 1-6, 2003.
- 20. Filip M, Frankowska M, Sadakierska-Chudy A, Suder A, Szumiec L, Mierzejewski P, Bienkowski P, Przegaliinski E, Cryan JF. GABA-B receptors as a therapeutic strategy in substance use disorders: focus on positive allosteric modulators. Neuropharmacol 2014 [epub ahead of print]
- 21. Franklin TR, Harper D, Kampman K, Kildea-McCree S, Jens W, Lynch KG, O'Brien CP, Childress AR. The GABA-B agonist baclofen reduces cigaretter consumption in a preliminary double-blind placebo-controlled smoking reduction study. Drug Alcohol Depend. 103: 30-36, 2009.
- 22. Franklin TR, Wang A, Sciortino N, Harper D, Li Y, Hakun J, Kildea S, Kampman K, Ehrman R, Detre JA, O'Brien CP and Childress AR. Modulation of resting brain cerebral blood flow by the Gaba B agonist, baclofen: a longitudinal perfusion fMRI study. Drug Alcohol Depend. 2011; 117: 176-183.
- 23. Galeotti N, Ghelardini C and Bartolini A. Piracetam and aniracetam antagonism of centrally active drug-induced antinociception. Pharm Biochm Behav 53: 943-950, 1996
- 24. Gordon NC, Gear RW, Heller PH, Paul S,, Miaskowski C and Levine JD. Enhancement of morphine analgesia by the GABA B agoinist baclofen. Neuroscience 69: 345-349, 1995
- 25. Gorsane M-A, Kebir O, Hache G, Blecha L, Aubin H-J, Reynaud M and Benyamina A. Is baclofen a revolutionary medication in alcohol addiction management? Review and recent updates. Substance Abuse 33: 336-349, 2012

- 26. Harmer JP and Larson BS. Pain relief from baclofen analgesia in a neuropathic pain patient who failed opioid and pharmacotherapy: case report J Pain Palliat Care Pharmacother 16: 61-64, 2002.
- 27. Heinrichs SC, Leite-Morris KA, Carey RJ, Kaplan GB. Baclofen enhances extinction of opiate conditioned place preference. Behav Brain Res. 207: 353-359, 2010.
- 28. Houston AJ, Wong JC, Ebenezer IS. A study on the involvement of GABA-B receptor ligands in stress-induced antinociception in male mice. Methods Find Exp Clin Pharmacol. 19: 167-171, 1997.
- 29. Ignatov IuD and Andreev BV. Role of opioid and adrenergic mechanisms in the analgesic action of the GABA-positive drugs. Biull Eksp Biol Med 105: 556-558, 1988.
- 30. Jasmin L, Rabkin SD, Granato A, Boudah A and Ohara PT. Analgesia and hyperalgesia from GABA-mediated modulation of the cerebral cortex. Nature 424: 316-320, 2003
- 31. Johnson BA, Swift RM, Addolorato G, Ciraulo DA, Myrick H. Safety and efficacy of GABA-ergic medications for treating alcoholism. Alcohol Clin Exp Res 29: 248-254, 2005.
- 32. Knisely JS, Wunsch MJ, Cropsey KL and Campbell ED. Presciption Opioid Misuse Index: a brief questionnaire to assess misuse. J Sub Abuse Treat 35: 380-386, 2008.
- 33. Knotkova H, Pappagallo M. Adjuvant analgesics. Med Clin North Am. 91: 113-124, 2007.
- 34. Kumar K, Sharma S, Kumar P, Deshmukh R. Therapeuti potential of GABA(B) receptor ligands in drug addiction, anxiety, depression and other CNS disorders. Pharmacol Biochem Behav 110: 174-184, 2013.
- 35. Leggio L, Garbutt JC, Addolorato G. Effectiveness and safety of baclofen in the treatment of alcohol dependent patients. CNS Neurol Disord Drug Targets 9: 33-44, 2010.
- 36. Leung NY, Whyle IM and Isbister GK. Baclofen overdose: defining the spectrum of toxicitiy. Emerg Med Australias. 18: 77-82, 2006.
- 37. Lim CR, Garant DS and Gale K. GABA agonist induced analgesia elicited from the lateral preoptic area in the rat. Eur J Pharmacol 107: 91-04, 1984.
- 38. Ling W and Shoptaw S. Baclofen as a cocaine anti-craving medication: a preliminary clinical study Neuropsychopharmacology 18: 493-404, 1998.
- 39. Maccioni P and Colombo G. Role of the GABA-B receptor in alcohols seeking and drinking behavior. Alcohol 43: 555-558, 2009.
- 40. Malcangio M and Bowery NG. Spinal cord SP release and hyperalgesia in monoarthritic rats: involvement of the GABA B receptor systems. Br. J Pharmacol. 113: 1561-1566, 1994.
- 41. Margetis K, Papagegeorgiou G, Gatzonis S, Politis K, Siatourni A and Sakas D. Intrathecal baclofen improves psychiatric symptoms in spasticity patients. J Clin Psychopharmacol 34: 374-379, 2014
- 42. Meng S, Quan W, Qi X, Su Z, Yang S. Effect of baclofen on morphine-induced conditioned place preference, extinction, and stress-induced reinstatement in chronically stressed mice. Psychopharmacol 231: 27-36, 2014.
- 43. Merlin JS, Herbey I, Starrels JL, Kertesz SG, Saag MS and Ritchie CS. Aberrant drug-related behaviors: a qualitative analysis of medical record documentation inpatients referred to an HIV/Chronic Pain Pain. Pain Med. 2014
- 44. Naderi N, Shafaghi B, Khodayar MJ and Zarindast MR. Interaction between GABA-B amd CB1 receptors in spinal pain pathways in rat. Eur J Pharmacol 514: 159-164, 2005.
- 45. Panerai AE, Massei R, deSilva E, Sacerdote P, Monza G, Mantegazza P. Baclofen prolongs the analgesic effect of fentanyl in man. Br. J Anaesth 57: 954-955, 1985.
- 46. Paterson NE, Froesti W, Markou A. The GABA-B receptor agonists baclofen and CGP44532 decreased nicotine self-administration in the rat. Psychopharmacol (Berl) 172: 179-186, 2003.

- 47. Porrino LJ, Hampson RE, Opris I and Deadwyler SA. Acute cocaine induced deficits in cognitive performance in rhesus macaque monkeys treated with baclofen. Psychopharmacol (Berl) 225: 105-114, 2013
- 48. Przesmycki K, Dzieciuch J and Kleinrok Z. The influence of GABA-ergic system on clonidine analgesia in rats. Pol J Pharmacol 46: 409-415, 1994.
- 49. Ramshini E, Alaei H, Reisi P, Alaei S and Shahidani S. The role of GABA B receptors in morphine self administration. In J Prev Med 4: 158-164, 2013.
- 50. Riahi E, Mirzaii-Dizgah I, Karimian SM, Roodsari HRS and Dehpour AR. Attenuation of morphine withdrawal signs by a GABA-B receptor agonist in the locus coeruleus of rats. Behaviroal Brain Res 196: 11-14, 2009.
- 51. Ross JC, Cook AM, Stewart GL and Fahy BG. Acute intratheecal baclofen withdrawal: a brief review of treatment options. Neurocrit Care 14: 103-108, 2011.
- 52. Roy CW and Wakefield IR. Baclofen pseudopsychosis: case report. Paraplegia 24: 318-321, 1986.
- 53. Sharma R, Mathur R and Nayar U. GABA B mediated analgesia in tonic pain in monkeys. Indian J Physiol Pharmacol 37: 189-193, 1993.
- 54. Silva JR, Silva ML and Prado WA. Analgesia induced by 2- or 100-Hz electroacupuncture in the rat tail-flick test depends on the activation of different descending pain inhibitory mechanisms. J. Pain 12: 51-60, 2011
- 55. Silversides JA and Scott KC. Diaete insipidus following overdose of baclofen and quetiapine. Anaesth Intensive Care 37: 319-320, 2009.
- 56. Spano MS, Fattore L, Fratta W, Fadda P. The GABA-B receptor agonist baclofen prevents heoin-induced reinstatement of heroin-seeking behavior in rats. Neuropharmacology 52: 1555-1562, 2007
- 57. Srivasta S, Hoon A, Ogborn J and Johnsont M. Acute onset rhythmic hiccup-like respirations secondary to oral baclofen toxicity. Pediat Neurol 51: 252-254, 2014.
- 58. Taira T, Kawamura H, Tanikawa T, Kawabatake H, Iseki H, Ueda A, Takakura K. A new approach to the control of central deafferentation pain spinal intrathecal baclofen. Acta Neurochir Suppl 64: 136-138, 1995.
- 59. Takeda M, Tanimoto T, Ikeda M, Kadoi J and Matsumoto S. Activation of GABA-B receptor inhibits the excitability of rat small diameter trigeminal root ganglion neurons. Neuroscience 123: 491-505, 2004.
- 60. Tamayo L, Rifo J and Contreras E. Influence of adrenergic and cholinergic mechanisms in baclofen induced analgesia. Gen Pharmacol 19: 87-89, 1988.
- 61. Tambeli, Levine JD, Gear RW. Centralization of noxious stimulus-induced analgesia (NSIA) is related to activity at inhibitiory synapses in the spinal cord. Pain 143: 228-232, 2009.
- 62. Terrence CF, Fromm GH and Tenicela R. Baclofen as an analgesic in chroinic peripheral nerve disease. Eur Neurol 24: 380-385, 1985.
- 63. Thomas DA, McGowan MK and Hammond DL. Microinjection of baclofen in the ventromedial medulla of rats: antinociception at low doses and hyperalgesia at high doses. J. Pharm Exp Therapeut 275: 274-284, 1995.
- 64. Tokuyama S, Takahashi M and Kaneto H. Participation of GABAergic systems in the production of antinociception by various stresses in mice. Japa J Pharmacol 60: 105-110, 1992.
- 65. Tyacke RJ, Lingford-Hughes A, Reed LJ and Nutt DJ. GABA-B receptors in addiction and its treatment. Adv. Pharmacol 58: 373-396, 2010.
- 66. Villas Boas GR, Zamboni CG, Peretti MC, Correia D, Rueda AV, Camarini R, Brunialti-Godard AL, and Boerngen-Lacerda R. Gaba(B) receptor agonist only reduces ethanol drinking in light-drinking mice. Pharmacol. Biochem Behav 102: 233-240, 2012.

- 67. Voigt R, Herrold AA and Napier TC. Baclofen facilitates the extinction of methamphetamine-iniduced conditioned place preference in rats. Behav Neurosci. 125: 261-267, 2011.
- 68. Vuittonet CL, Halse M, Leggio L, Fricchione SB, Brickley M, Haass-Koffler CL, Tavares T, Swift RM and Kenna GA. Pharmacotherapy for alcoholic patients with alcoholic liver disease. Am J Health Syst Pharm 71: 1265-1276, 2014.
- 69. Xiao W, Naso L and Bennett GJ. Experimental studies of potential analgesics for the treatment of chemotherapy-evoked painful neuropathies. Pain Med 9:505-517, 2008.
- 70. Yang K AND Ma H. Blockade of GABA(B) receptiors facilitates evoked neurotransmitter release at spinal dorsal horn synapse. Neuroscience 193: 411-420, 2011.
- 71. Zarrindast MR and Djavdan M. GABA-A-antagonists and baclofen analgesia. Gen Pharmacol 19: 703-706, 1988
- 72. Zharrindast MR, Khodjastehfar E, Oryan S, Torkaman-Boutorabi A. Baclofen-impairment of memory retention in rats: possible interaction with adrenoceptor mechanism(s) Eur J Pharmacol 411: 283-286, 2001.